CLINICAL TRIAL: NCT02701348
Title: Radiological and Biological Tumoural and Peri-tumoural Factors in Neoadjuvant Endocrine-treated Breast Cancers
Acronym: BARONET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Tayside (Other Government)
Responsible Party: Principal Investigator, Jane MacAskill, Dr. Jane MacAskill, NHS Tayside
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2015ON09
Record Dates: First submitted 2015-12-15; First posted 2016-03-08 (Estimated); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Breast Cancer
Keywords: neoadjuvant endocrine
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole; Aromatase Inhibitors; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Shearwave elastography — Patients with primary breast cancer receiving neoadjuvant letrozole will undergo radiological assessment with digital mammogram, ultrasound (US) including shearwave elastography (SWE). These will be performed at 3 monthly intervals until surgical intervention is considered feasible.
Drug: Letrozole — Patients will be receiving neoadjuvant letrozole as standard therapy for breast cancer
  Other Names: Aromatase inhibitor
Procedure: Breast core biopsy — Core biopsies will be taken at diagnosis, and at the time of surgery to allow biological assessment of changes in tumour
Other: Magnetic Resonance Imaging — Breast MRI scans will be performed at time of diagnosis and prior to surgery to allow comparison of MRI change and response to treatment

SUMMARY:
The purpose of this study is to monitor the change in cancer size in women with breast cancer on anti-hormone treatment using different types of assessment including ultrasound scan (US), shearwave elastography (SWE) and magnetic resonance imaging (MRI), and assess how this corresponds to the changes in the cancer biology.

DETAILED DESCRIPTION:
Background Endocrine resistance is a significant problem in the management of breast cancer, with increasing evidence that the tumour microenvironment is influential on tumour growth and disease resistance. The neoadjuvant setting provides an excellent opportunity to observe tumour response to treatment in vivo, allowing development of methods for monitoring and predicting response to treatment.

Aims To assess potential radiological and biological tumoural and peri-tumoural biomarkers in patients before and during neoadjuvant endocrine treatment. Our hypothesis is that there will be less response in women with abnormal peri-tumoural stroma, and that tumours with high monocarboxyl transporter (MCT4) and loss of caveolin-1 in stroma are resistant to endocrine treatment.

Techniques and Methodology Patients with primary breast cancer receiving neoadjuvant letrozole will undergo radiological assessment with digital mammogram, US including SWE, and MRI. Core biopsies will be taken at diagnosis and at surgery from tumour and peri-tumoural stroma, and assessed for biomarkers lysyl oxidase (LOX), fibronectin, collagen, proliferation, MCT4 and caveolin-1. All data will be correlated to peri-tumoural abnormalities on MRI and SWE.

Impact on breast cancer research This study will provide information on the ability of SWE and MRI to predict and detect endocrine resistance, correlated with biological markers that are associated with endocrine resistance. Identifying resistant tumours can prevent unnecessary treatment and reduce risks of recurrence as alternative or additional therapies can be utilised.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women: Defined as >12 months amenorrhoea in absence of medical therapy known to induce this; or bilateral oophorectomy; or if last menses <12 months before starting treatment, FSH >35 IU/L and LH >40 IU/L.
* ER positive (Allred score >3) invasive breast cancer
* Staging as T1-4, N0-2, M0
* Patient agreed to neoadjuvant endocrine therapy as recommended by MDT
* Fresh tissue stored at time of diagnostic core biopsy
* Suitable for, and tolerant of MRI scan
* Fit for surgical intervention at time of entry into study

Exclusion Criteria:

* Premenopausal or unable to determine menopausal status
* Not fit for surgical intervention due to co-morbidities
* Contraindication for MRI (including severe claustrophobia)
* Current use of HRT, or HRT use at time of diagnostic core biopsy

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-05; Primary Completion 2020-12-24 (Actual); Study Completion 2020-12-24 (Actual)

PRIMARY OUTCOMES:
Change in Proliferative response | At surgery, min 3 months max 24 months
  Pathological response to treatment by proliferation (Ki67) (%)
Change in Pathological response | At surgery, min 3 months max 24 months
  Residual cancer burden score
Change in Shearwave stiffness | 0,3,6, up to 24 months
  shearwave stiffness (kPa)

SECONDARY OUTCOMES:
Change in peritumoural imaging on MRI | 0 months and surgery (min 3 months, max 24 months)
  MRI - digital contrast enhanced (DCE) and diffusion weighted imaging (DWI)
caveolin-1 | 0 months and at time of surgery (min 3 months, max 24 months)
  peri-tumoural immunohistochemical analysis
Monocarboxyl transport 4 | 0 months and at time of surgery (min 3 months, max 24 months)
  peri-tumoural immunohistochemical analysis
lysyl oxidase | 0 months and at time of surgery (min 3 months, max 24 months)
  peri-tumoural immunohistochemical analysis
fibronectin | 0 months and at time of surgery (min 3 months, max 24 months)
  peri-tumoural immunohistochemical analysis
collagen | 0 months and at time of surgery (min 3 months, max 24 months)
  peri-tumoural immunohistochemical analysis

CONTACTS AND LOCATIONS:
Overall Officials: E. Jane Macaskill, MBChB, MD, FRCSEd, Principal Investigator — NHS Tayside
Locations (1):
- Stefani Clinical Trials Unit, Ninewells Hospital and Medical School, Dundee, Angus, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No individual data sharing